CLINICAL TRIAL: NCT05525351
Title: The Application and Validation of Triple Drug Response Surface Models on Density Spectral Array in Clinical Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-02-019B
Record Dates: First submitted 2022-08-11; First posted 2022-09-01 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia; Drug Interaction; Anesthesia; Functional
Keywords: Three-drug response surface model; Thoracic surgery; Bispectral index; Patient state index; propofol; dexmedetomidine; opioid
MeSH Terms: interventions — Propofol; Alfentanil; Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- NI-VATS (Non-intubated video-assisted thoracoscopic surgery): This is a purely observational study of the routine anesthetic practice involving the simultaneous use of three drugs. Types of surgery (non-intubated video-assisted thoracoscopic surgery or video-assisted thoracoscopic surgery) are discussed and decided totally by patients and surgeons independently.
  NI-VATS: induction and maintenance are achieved by propofol, alfentanil and dexmedetomidine. Patients are monitored with standard monitors (electrocardiography, Non-invasive blood pressure, and pulse oximetry), arterial blood pressure (ABP) and bispectral index (BIS) or Patient State Index (PSI) monitor. Patients are observed in the recovery unit with designate nursing staff until full conscious recovery before discharge.
  Interventions: Device: Bispectral index (BIS) or Patient State Index (PSI); Drug: Propofol; Drug: Alfentanil; Drug: Dexmedetomidine
- VATS (video-assisted thoracoscopic surgery): This is a purely observational study of the routine anesthetic practice involving the simultaneous use of three drugs. Types of surgery (non-intubated video-assisted thoracoscopic surgery or video-assisted thoracoscopic surgery) are discussed and decided totally by patients and surgeons independently.
  NI-VATS: induction and maintenance are achieved by propofol, alfentanil and dexmedetomidine. Patients are monitored with standard monitors (electrocardiography, Non-invasive blood pressure, and pulse oximetry), arterial blood pressure (ABP) and bispectral index (BIS) or Patient State Index (PSI) monitor. Patients are observed in the recovery unit with designate nursing staff until full conscious recovery before discharge.
  Interventions: Device: Bispectral index (BIS) or Patient State Index (PSI); Drug: Propofol; Drug: Alfentanil; Drug: Dexmedetomidine

INTERVENTIONS:
Device: Bispectral index (BIS) or Patient State Index (PSI) — After giving routine anesthetic medications, the investigators assess the depth of anesthesia based on bispectral index (BIS) or Patient State Index (PSI). BIS is maintained between 40 - 60 and PSI between 25 - 50. The vital signs, BIS or PSI are recorded automatically and continuously through computerized software. Upon conclusion of the surgery or examination, the patient is observed until return of consciousness (MOAA/S = 5) before sending them to the recovery unit.
Drug: Propofol — The investigators assess the depth of anesthesia based on bispectral index (BIS) or Patient State Index (PSI) after routine drug regimen is given. BIS is maintained between 40 and 60 and or PSI between 25 and 50. The drug doses are given as a part of routine anesthesia practice and is identical regardless of study participation. Propofol is given via target control pump with typical target effect-site propofol concentration 1-5 ug/mL according to patient condition, BIS or PSI value and DSA. The timing and doses are recorded for backend analysis. At the conclusion of the surgery or examination, the patient is observed in the surgery or examination room until return of consciousness before sending them to the recovery unit.
Drug: Alfentanil — The investigators assess the depth of anesthesia based on bispectral index (BIS) or Patient State Index (PSI) after routine drug regimen is given. BIS is maintained between 40 and 60 and or PSI between 25 and 50. The drug doses are given as a part of routine anesthesia practice and is identical regardless of study participation. Typical alfentanil ranged from 0~1000mcg according to patient condition, BIS or PSI value and DSA. The timing and doses are recorded for backend analysis. At the conclusion of the surgery or examination, the patient is observed in the surgery or examination room until return of consciousness before sending them to the recovery unit.
Drug: Dexmedetomidine — The investigators assess the depth of anesthesia based on bispectral index (BIS) or Patient State Index (PSI) after routine drug regimen is given. BIS is maintained between 40 and 60 and or PSI between 25 and 50. The drug doses are given as a part of routine anesthesia practice and is identical regardless of study participation. Typical Dexmedetomidine ranged from 0.5-1 ug/kg/hr according to patient condition, BIS or PSI value and DSA. The timing and doses are recorded for backend analysis. At the conclusion of the surgery or examination, the patient is observed in the surgery or examination room until return of consciousness before sending them to the recovery unit.

SUMMARY:
Precision anesthesia is the current trend. The benefits including faster recovery, earlier return to normal activity, increased patient satisfaction and shorter length of stay. In order to avoid unnecessarily deep or too light anesthesia, processed electroencephalogram (EEG) monitors are applied for accurate assessment of the depth of anesthesia (DoA). Bispectral index (BIS) and PSI monitor are among the most widely used. Recently, density spectral array (DSA) has been developed to facilitate the interpretation of EEG signals. Real-time DSA EEG monitoring helps in detecting even subtle changes in the depth of anesthesia and provides more comprehensive information then simple digits.

An emerging field of pharmacodynamics in anesthesia is the response surface models. They describe the interaction of different anesthetics during sedation or anesthesia. Our research team has developed the first comprehensive two-drug response surface models for midazolam and alfentanil during gastrointestinal procedural sedations. However, adequate anesthesia is often achieved with multiple drugs. Two-drug models thus have limited applications. We aim to extend the models into three-drug interactions where it can be used for a broader range of clinical scenarios.

The main goal of the study is to establish and validate the three-drug response surface model by collecting and analyzing EEG parameters (BIS or PSI values, DSA, SEF95 (95% spectral edge frequency) and MF (Median frequency) ) from 60 patients undergoing general anesthesia for thoracic surgeries. We aim to establish the models that help anesthesiologist to achieve rapid emergence, appropriate analgesia, adequate DoA, and patient safety. The secondary aim is to apply this model to provide a guideline for drug dosage adjustment and improve the quality of anesthesia.

DETAILED DESCRIPTION:
This is an observational study of the routine clinical practice of anesthesia and surgery with no specific additional interventions required. Types of surgery (non-intubated video-assisted thoracoscopic surgery or video-assisted thoracoscopic surgery) are discussed and decided totally by patients and surgeons.

Data acquisition (Non-intubated video-assisted thoracoscopic surgery, NI-VATS)

1. After screening for eligible patients, protocol and study details will be thoroughly explained to them.
2. Each patient received standard anesthetic care of our institute. Strict fasting protocols were followed. A 22 or 20-gauge intravenous catheter was secured for drug administration.

   Monitors are comprised of ECG (electrocardiography), oxygenation saturation (SpO2) ,NIBP (non-invasive blood pressure)and arterial blood pressure (ABP). ECG, SpO2 and ABP were monitored continuously and NIBP were measured every 60 minutes. Supplemental oxygen was given via high flow nasal cannula, and SpO2 (oxygenation saturation) maintained above 90%. Induction and maintenance of anesthesia is achieved by intravenous propofol, dexmedetomidine and alfentanil. Dosage are according to anesthesiologist's preference. Anesthetic depth was monitored with BIS or PSI monitor.
3. BIS or PSI monitor is continuously recorded throughout the surgery to collect EEG parameters such as BIS or PSI values, DSA, SEF95 (95% spectral edge frequency) and MF (Median frequency). MOAA/S score would be recorded at induction and emergence phase.
4. At the end of the procedure, the patient was observed until return of consciousness (MOAA/S > 5). Collected data will be randomly divided into a model training group and a validation group after data acquisition by computer randomization using computer clock as seed.

Data acquisition (Video-assisted thoracoscopic surgery, VATS)

1. After screening for eligible patients, protocol and study details will be thoroughly explained to them.
2. Each patient received standard anesthetic care of our institute. Strict fasting protocols were followed. A 22 or 20-gauge intravenous catheter was secured for drug administration. Monitors are comprised of ECG (electrocardiography), oxygenation saturation (SpO2) ,NIBP (non-invasive blood pressure)and arterial blood pressure (ABP). ECG, SpO2 and ABP were monitored continuously and NIBP were measured every 60 minutes. Induction and maintenance of anesthesia is achieved by intravenous propofol, dexmedetomidine, alfentanil and neuromuscular blocking agents. Dosage are according to anesthesiologist's preference. Anesthetic depth was monitored with BIS or PSI.
3. After double lumen endotracheal tube placement, FiO2: 100 % and fresh gas flow at 1~6 L/m was set. BIS or PSI monitor is continuously recorded throughout the surgery to collect EEG parameters such as BIS or PSI values, DSA, SEF95 (95% spectral edge frequency) and MF (Median frequency). MOAA/S score would be recorded at induction and emergence phase
4. At the end of the procedure, endotracheal tube was removed if the patient was breathing smoothly. The patient was observed until return of consciousness (MOAA/S > 5). Collected data will be randomly divided into a model training group and a validation group after data acquisition by computer randomization using computer clock as seed.

Model building, assessment and validation (both groups)

1. Collected data were fed to a pharmacokinetic simulation software (TIVA trainer Version 9.1) to calculate second-by-second plasma and effect-site drug concentration changes for all three drugs. The training patient group is used for model training. The bootstrap technique is used with 2000 iterations. Model fit was optimized using -2 Log likelihood (-2LL).
2. MOAA/S, BIS or PSI models would be constructed.
3. The results are validated with the validation patient data to confirm its clinical utility.

Receiver operating characteristics (ROC) curve analysis is used to assess the quality of model prediction. ROC and area under the curve (AUC) will be compared between the training and validation group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 85
* Scheduled for Non-intubated VATS or VATS surgery depending on study arm.
* American Society of Anesthesiologists (ASA) physical status I to III.

Exclusion Criteria:

* hearing impairment
* neurologic or behavioral disorders
* habitual sedative use
* alcoholism
* allergy to dexmedetomidine, alfentanil or propofol
* resting room air SpO2 < 90%.
* History of upper airway tumors

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NI-VATS (non-intubated Video-Assisted Thoracic Surgery) population: The investigators plan to enroll patients who will receive NI-VATS under general anesthesia. These patients will be screened for eligibility.
  VATS (Video-Assisted Thoracic Surgery) population: The investigators plan to enroll patients who will receive VATS under general anesthesia. These patients will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Bispectral index (BIS) value or Patient state index (PSI) value | EEG are recorded starting from anesthesia induction, and stopped after emergence when surgery ends as a part of routine anesthesia.
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. The recorded BIS or PSI value reading is uniform and contains only a unitless number ranging from 0 to 100. Different procedures do not give different units. These values are part of anesthetic depth evaluation and the recordings are aggregated to perform fit in a mathematic model.
EEG frequency | EEG are recorded starting from anesthesia induction, and stopped after emergence when surgery ends as a part of routine anesthesia.
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. Raw EEG data are recorded and analyzed afterwards. Spectral analysis of the alpha, beta, gamma, theta and delta features will be performed. Individual band powers are summed separately. EEG frequency will be recorded continuously during the total anesthesia time to perform fit in a mathematic model.
Power of the EEG signal | EEG are recorded starting from anesthesia induction, and stopped after emergence when surgery ends as a part of routine anesthesia.
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. Raw EEG data are recorded and analyzed afterwards. Spectral analysis of the alpha, beta, gamma, theta and delta features will be performed. Individual band powers are summed separately. Power of the EEG signal represents amount of activity in certain frequency bands. Power of the EEG signal will be recorded continuously during the total anesthesia time to perform fit in a mathematic model.
Spectral edge frequency 90 (SEF 90) | EEG are recorded starting from anesthesia induction, and stopped after emergence when surgery ends as a part of routine anesthesia.
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. Raw EEG data are recorded and analyzed afterwards. Spectral analysis of the alpha, beta, gamma, theta and delta features will be performed. Individual band powers are summed separately. Spectral edge frequency 90 (SEF 90) represents the frequency below which 90 % of the EEG power is located. SEF 90 will be recorded continuously during the total anesthesia time to perform fit in a mathematic model.
Median frequency (MF) | EEG are recorded starting from anesthesia induction, and stopped after emergence when surgery ends as a part of routine anesthesia
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. Raw EEG data are recorded and analyzed afterwards. Spectral analysis of the alpha, beta, gamma, theta and delta features will be performed. Individual band powers are summed separately. The median frequency represents the frequency below and above which lies 50% of the total power in the EEG. MF will be recorded continuously during the total anesthesia time to perform fit in a mathematic model.

SECONDARY OUTCOMES:
Modified Observer's Assessment Alertness Scale(MOAA/S) score | MOAA/S score will be recorded specifically at induction and emergence phase
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. MOAA/S is a unitless score between 0 and 5 and is applicable in different anesthesia settings. Different procedures do not give different MOAA/S units. Return of consciousness is defined by a score of MOAA/S greater than 4. The score is a part of anesthetic depth evaluation and the recordings are aggregated to perform fit in a mathematic model.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Yung Tsou, MD. PhD., Study Director — Taipei Veterans General Hospital; National Yang-Ming University
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liou JY, Ting CK, Teng WN, Mandell MS, Tsou MY. Adaptation of non-linear mixed amount with zero amount response surface model for analysis of concentration-dependent synergism and safety with midazolam, alfentanil, and propofol sedation. Br J Anaesth. 2018 Jun;120(6):1209-1218. doi: 10.1016/j.bja.2018.01.041. Epub 2018 Apr 17. PMID 29793588
- [Background] Liou JY, Ting CK, Mandell MS, Chang KY, Teng WN, Huang YY, Tsou MY. Predicting the Best Fit: A Comparison of Response Surface Models for Midazolam and Alfentanil Sedation in Procedures With Varying Stimulation. Anesth Analg. 2016 Aug;123(2):299-308. doi: 10.1213/ANE.0000000000001299. PMID 27192475
- [Background] LaPierre CD, Johnson KB, Randall BR, Egan TD. A simulation study of common propofol and propofol-opioid dosing regimens for upper endoscopy: implications on the time course of recovery. Anesthesiology. 2012 Aug;117(2):252-62. doi: 10.1097/ALN.0b013e31825fb1b2. PMID 22728781
- [Background] Ting CK, Johnson KB, Teng WN, Synoid ND, Lapierre C, Yu L, Westenskow DR. Response surface model predictions of wake-up time during scoliosis surgery. Anesth Analg. 2014 Mar;118(3):546-53. doi: 10.1213/ANE.0000000000000094. PMID 24557102
- [Background] Liou JY, Ting CK, Huang YY, Tsou MY. Previously published midazolam-alfentanil response surface model cannot predict patient response well in gastrointestinal endoscopy sedation. J Chin Med Assoc. 2016 Mar;79(3):146-51. doi: 10.1016/j.jcma.2015.11.002. Epub 2016 Jan 28. PMID 26831450
- [Background] [40 years of scientific-research work in medicine]. Patol Fiziol Eksp Ter. 1969 May-Jun;13(3):91-4. No abstract available. Russian. PMID 4907643
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] de Heer IJ, Bouman SJM, Weber F. Electroencephalographic (EEG) density spectral array monitoring in children during sevoflurane anaesthesia: a prospective observational study. Anaesthesia. 2019 Jan;74(1):45-50. doi: 10.1111/anae.14458. Epub 2018 Oct 27. PMID 30367683